CLINICAL TRIAL: NCT04860206
Title: Vpliv COVID19 na Izgubo Funkcionalnih zmožnosti Pacientov po zaključenem bolnišničnem Zdravljenju The Effect of COVID19 on the Loss of Functional Capacity of Patients After Hospitalization
Brief Title: Post COVID19 Functional and Cognitive Assessments
Acronym: PostCovidZRS
Status: Completed | Type: Observational
Sponsor: Science and Research Centre Koper (Other)
Collaborators: Hospital of Izola (Unknown); University of Trieste (Other); University of Padova (Other); University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: PC-ZRS-SBI
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Covid19; Respiratory Disease; Walking, Difficulty; Cognitive Decline
Keywords: COVID19; functional outcomes; respiratory function
MeSH Terms: conditions — COVID-19; Respiration Disorders; Mobility Limitation; Cognitive Dysfunction; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the proposed study is to evaluate the impact of coronavirus (2019-nCoV), hereafter COVID -19, on patients' loss of functional capacity after completion of hospital treatment. Specifically, the research will focus on examining changes in musculoskeletal, cardiovascular, and respiratory function, as well as motor control. In addition, we aim to evaluate rehabilitation treatments after recovery from COVID -19 and consider additional preventive measures based on previous experience.

DETAILED DESCRIPTION:
The combination of such a severe respiratory disease as COVID -19 with motor inactivity could have very serious consequences for a person's general health even after COVID -19 symptoms have subsided. To date, the effects of COVID -19 on individual muscle status have not been extensively studied. Therefore, the main objective of this study will be to evaluate the muscle status of patients after COVID -19. In addition, we will be interested in longitudinal monitoring of individuals' rehabilitation, where they will receive instructions based on measured outcomes at hospital discharge. We will also be interested in considering additional preventive measures for future patients based on previous experience of infected and hospitalized COVID -19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Completed hospital treatment after a positive COVID-19 test
* Signed written consent

Exclusion Criteria:

* Still testing positive for COVID -19 at discharge.
* Severe musculoskeletal injuries (e.g., disability).
* Inability to follow instructions when performing the test.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All male and female patients who tested positive for COVID -19 and were discharged from hospital care will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | Change in time on TUG between both assessment points (pre- to 2 months post-measurement)
  Functional performance of the patients from sitting to standing, walking and turning
Pulse wave velocity (PWV) | Change in PWV between both assessment points (pre- to 2 months post-measurement)
  Measuring endothelium function in supine
Spirometry | Change in FVC (%) between both assessment points (pre- to 2 months post-measurement)
  Measurement of lung function, specifically the forced vital capacity (FVC)

SECONDARY OUTCOMES:
Walking velocity | Change in gait velocity between both assessment points (pre- to 2 months post-measurement)
  measurement of gait velocity on the 4m path.
Trail making test B | Change in time to solve the TMT B test between both assessment points (pre- to 2 months post-measurement)
  Measurement of executive control using the TMT B test

CONTACTS AND LOCATIONS:
Locations (1):
- SB Izola, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ammar A, Chtourou H, Boukhris O, Trabelsi K, Masmoudi L, Brach M, Bouaziz B, Bentlage E, How D, Ahmed M, Mueller P, Mueller N, Hsouna H, Aloui A, Hammouda O, Paineiras-Domingos LL, Braakman-Jansen A, Wrede C, Bastoni S, Pernambuco CS, Mataruna L, Taheri M, Irandoust K, Khacharem A, Bragazzi NL, Strahler J, Washif JA, Andreeva A, Khoshnami SC, Samara E, Zisi V, Sankar P, Ahmed WN, Romdhani M, Delhey J, Bailey SJ, Bott NT, Gargouri F, Chaari L, Batatia H, Ali GM, Abdelkarim O, Jarraya M, Abed KE, Souissi N, Gemert-Pijnen LV, Riemann BL, Riemann L, Moalla W, Gomez-Raja J, Epstein M, Sanderman R, Schulz S, Jerg A, Al-Horani R, Mansi T, Jmail M, Barbosa F, Ferreira-Santos F, Simunic B, Pisot R, Pisot S, Gaggioli A, Zmijewski P, Apfelbacher C, Steinacker J, Saad HB, Glenn JM, Chamari K, Driss T, Hoekelmann A, On Behalf Of The Eclb-Covid Consortium. COVID-19 Home Confinement Negatively Impacts Social Participation and Life Satisfaction: A Worldwide Multicenter Study. Int J Environ Res Public Health. 2020 Aug 27;17(17):6237. doi: 10.3390/ijerph17176237. PMID 32867287
- [Background] Ammar A, Brach M, Trabelsi K, Chtourou H, Boukhris O, Masmoudi L, Bouaziz B, Bentlage E, How D, Ahmed M, Muller P, Muller N, Aloui A, Hammouda O, Paineiras-Domingos LL, Braakman-Jansen A, Wrede C, Bastoni S, Pernambuco CS, Mataruna L, Taheri M, Irandoust K, Khacharem A, Bragazzi NL, Chamari K, Glenn JM, Bott NT, Gargouri F, Chaari L, Batatia H, Ali GM, Abdelkarim O, Jarraya M, Abed KE, Souissi N, Van Gemert-Pijnen L, Riemann BL, Riemann L, Moalla W, Gomez-Raja J, Epstein M, Sanderman R, Schulz SV, Jerg A, Al-Horani R, Mansi T, Jmail M, Barbosa F, Ferreira-Santos F, Simunic B, Pisot R, Gaggioli A, Bailey SJ, Steinacker JM, Driss T, Hoekelmann A. Effects of COVID-19 Home Confinement on Eating Behaviour and Physical Activity: Results of the ECLB-COVID19 International Online Survey. Nutrients. 2020 May 28;12(6):1583. doi: 10.3390/nu12061583. PMID 32481594
- [Background] Pisot R, Marusic U, Biolo G, Mazzucco S, Lazzer S, Grassi B, Reggiani C, Toniolo L, di Prampero PE, Passaro A, Narici M, Mohammed S, Rittweger J, Gasparini M, Gabrijelcic Blenkus M, Simunic B. Greater loss in muscle mass and function but smaller metabolic alterations in older compared with younger men following 2 wk of bed rest and recovery. J Appl Physiol (1985). 2016 Apr 15;120(8):922-9. doi: 10.1152/japplphysiol.00858.2015. Epub 2016 Jan 28. PMID 26823343